CLINICAL TRIAL: NCT06843902
Title: ImproviNg Coronary Vascular Health in Women With Risk Factors fOR Myocardial Infarction Type 2 (INFORM-2)
Brief Title: Improving Coronary Vascular Health in Women
Acronym: INFORM_2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Markella V. Zanni,M.D., Associate Professor of Medicine, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024P001952; R01HL170905 (NIH)
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: HIV-1-infection; Coronary Microvascular Dysfunction; Metabolic Disease
Keywords: HIV; women; diabetes; chronic kidney disease; SGLT2 inhibitor therapy; coronary flow reserve; cardiovascular disease prevention
MeSH Terms: conditions — Metabolic Diseases; Diabetes Mellitus; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Health education plus subspecialty clinic referral for consideration of SGLT2 inhibitor therapy (Experimental): Participants randomized to this study arm will receive health education and will be referred to establish clinical care in either the MGH Lipid and Metabolism Clinic or the MGH Renal Clinic for consideration of SGLT2 inhibitor therapy. By study design (inclusion criteria), participants will have a clinical indication for SGLT2 inhibitor therapy (either diabetes or chronic kidney disease). SGLT2 inhibitor therapy (e.g. empagliflozin 10 mg by mouth daily or dapagliflozin 10 mg by mouth daily) may or may not be prescribed by the subspecialty clinician as part of routine clinical care, according to the clinician's clinical judgement. Participants will also receive health education.
  Interventions: Other: Health Education
- Health Education (Other): Participants randomized to this study arm will receive health education alone.
  Interventions: Other: Health Education; Other: Subspecialty clinic referral

INTERVENTIONS:
Other: Health Education — Health Education
Other: Subspecialty clinic referral — This intervention will entail referred to establish clinical care in either the MGH Lipid and Metabolism Clinic or the MGH Renal Clinic for consideration of SGLT2 inhibitor therapy. SGLT2 inhibitor therapy (e.g. empagliflozin 10 mg by mouth daily or dapagliflozin 10 mg by mouth daily) may or may not be prescribed by the subspecialty clinician as part of routine clinical care, according to the clinician's clinical judgement.
  Arms: Health Education

SUMMARY:
Women with HIV have an increased risk of having a myocardial infarction (heart attack) as compared to women without HIV. One of the mechanisms underlying the increased risk of myocardial infarction among women with HIV may involve reduced ability to increase blood flow through large and small coronary arteries at times when increased flow of oxygen-carrying blood is needed. We are conducting a study randomizing women with HIV and either diabetes, chronic kidney disease, or both to health education alone or to health education plus referral to see either an Endocrinologist or a Nephrologist in a subspecialty clinic for consideration of treatment with medication in a class known as sodium glucose transporter 2 (SGLT2) inhibitors. SGLT2 inhibitors are clinically approved for use in patients with diabetes or chronic kidney disease but have been shown to be underutilized in people with HIV. One of our key analytic aims will be to test if SGLT2 inhibitor therapy results in improved blood flow through the large and small coronary arteries among women with HIV and either diabetes, chronic kidney disease, or both but who have no history of myocardial infarction. A second aim will be to test if subspecialty clinic referral (with or without SGLT2 inhibitor therapy prescription) results in improved blood flow through the large and small coronary arteries among the same group.

DETAILED DESCRIPTION:
Women with HIV have an increased risk of having a myocardial infarction (heart attack) as compared to women without HIV. One of the mechanisms underlying the increased risk of myocardial infarction among women with HIV may involve reduced ability to increase blood flow through large and small coronary arteries at times when increased flow of oxygen-carrying blood is needed. We are conducting a study randomizing women with HIV and either diabetes, chronic kidney disease, or both to health education alone or to health education plus referral to see either an Endocrinologist or a Nephrologist in a subspecialty clinic for consideration of treatment with medication in a class known as sodium glucose transporter 2 (SGLT2) inhibitors. SGLT2 inhibitors are clinically approved for use in patients with diabetes or chronic kidney disease but have been shown to be underutilized in people with HIV. Prior to randomization, to confirm eligibility, participants will have undergone history, physical, lab tests, and cardiac positron emission tomography/computed tomography (PET/CT) scanning to confirm that there is a measure of impairment in stimulated blood flow through the large and small arteries of the heart. Randomized participants in both groups will be followed for 6 months and then will undergo repeat history, physical, laboratory testing, and repeat cardiac PET/CT scanning. One of our key analytic aims will be to test if SGLT2 inhibitor therapy results in improved blood flow through the large and small coronary arteries among women with HIV and either diabetes, chronic kidney disease, or both but who have no history of myocardial infarction. A second aim will be to test if subspecialty clinic referral (with or without SGLT2 inhibitor therapy prescription) results in improved blood flow through the large and small coronary arteries among the same group. We will also investigate effects of SGLT inhibitor therapy (and, separately, of subspecialty clinic referral) on fat tissue around the heart, as well as on blood and urine-based markers of metabolic disease and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* female sex-at-birth
* self-report of HIV on stable antiretroviral therapy ≥180 days
* age 45 -75 years
* at least 1 of the following 3 conditions: i) type 2 diabetes mellitus ii) estimated glomerular filtration rate 30-60 ml/min/1.73 m2 iii) urine albumin to creatinine ratio >30 mg/g
* coronary flow reserve <2.5 or stress myocardial blood flow <2.5 on screening cardiac positron emission tomography/computed tomography

Exclusion Criteria:

* current SGLT2 inhibitor use
* known allergy to SGLT2 inhibitor use
* type 1 diabetes or ketoacidosis prone diabetes (diabetes with a history of ketoacidosis)
* self-reported history of polycystic kidney disease
* self-reported history of myocardial infarction, stroke, or coronary revascularization
* stable or unstable angina
* self-reported history of heart failure
* hemoglobin A1c ≥8.5% at screen
* uncontrolled hypertension at screen, defined as systolic blood pressure ≥180 mm Hg and/or diastolic blood pressure ≥110 mm Hg
* estimated glomerular filtration rate <30 ml/min/1.73 m2
* currently receiving hemodialysis or peritoneal dialysis
* CD4 <400 cell/mm3
* current treatment with systemic (oral, IV, IM or intra-articular) steroids or anti-inflammatory/immune suppressant therapies (excluding topical therapies, UV therapy, ASA-derivatives, or NSAIDs) for any indication, including kidney disease
* pregnancy or breastfeeding
* known allergy to 13N Ammonia/82Rubidium or to Regadenoson/Adenosine
* concurrent enrollment in conflicting research study
* self-reported history of recurrent urinary tract-infections (≥2 urinary tract infections within 6 months or ≥3 within a year) and/or recurrent vaginal yeast infections (≥2 vaginal yeast infections within 6 months or ≥3 within a year)

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Coronary Flow Reserve | 24 weeks
  Change in coronary flow reserve by cardiac positron emission tomography
Ectopic Adipose Tissue | 24 weeks
  Change in ectopic adipose tissue reserve by cardiac computed tomography

SECONDARY OUTCOMES:
Kidney-related biomarkers | 24 weeks
  Urine and serum biomarkers related to kidney health and disease
Metabolic biomarkers | 24 weeks
  Urine and serum biomarkers relating to metabolism (including glucose and lipid metabolism)
Immune/inflammatory biomarkers | 24 weeks
  Urine and serum biomarkers relating to inflammation and immune activation
HIV-specific parameters | 24 weeks
  Serum variables relating to HIV disease (such as HIV-1 viral load, CD4 T cell count, CD8 T cell count)

CONTACTS AND LOCATIONS:
Overall Officials: Markella V Zanni, MD, Principal Investigator — MGH/HMS
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Plans are for IPD to be shared to the NIH BioLINCC data repository.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available 12 months after study completion and will remain available for a duration of time consonant with NIH policies.
Access Criteria: Access criteria are as per the NIH BioLINCC data repository.